CLINICAL TRIAL: NCT01362127
Title: Adjuvant Treatment of Cancer of the Esophagus or Cardia Before Resection With Curative Intent. Comparative Study Between Chemotherapy and Radiochemotherapy
Brief Title: Neoadjuvant Chemotherapy Versus Radiochemotherapy for Cancer of the Esophagus or Cardia
Acronym: NeoRes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: University Hospital, Umeå (Other); Region Örebro County (Other); Sahlgrenska University Hospital (Other); Ullevaal University Hospital (Other); Haukeland University Hospital (Other); Oslo University Hospital (Other); St. Olavs Hospital (Other); Malarhospital Eskilstuna (Unknown)
Responsible Party: Principal Investigator, Magnus Nilsson, Ass Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU-nr 2006-001785-16; 2006-001785-16 (EudraCT Number)
Record Dates: First submitted 2011-05-26; First posted 2011-05-27 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Carcinoma, Squamous Cell; Adenocarcinoma of the Esophagus and Gastric Cardia
Keywords: Histologically confirmed squamos cell carcinoma or adenocarcinoma of the esophagus and gastric cardia.Suitable for surgery.
MeSH Terms: conditions — Carcinoma, Squamous Cell; Adenocarcinoma Of Esophagus | interventions — Drug Therapy; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiochemotherapy (Active Comparator): Arm I: Radiochemotherapy + Surgery
  Interventions: Drug: Chemotherapy; Radiation: Radiochemotherapy
- Chemotherapy (Active Comparator): Arm II: Chemotherapy + surgery
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Cisplantin 100 mg/m2 day 1. 5-fluoracil 750 mg/m2/24 hours infusion day 1-5. Three cycles. In the chemoradiation arm the radiotherapy start week 4 and continuing until week 7. Dose adjustet according to current LPK and TPK values.
  Other Names: Suffering moderate/severe hearing impairment and/or tinnitus cisplatin can be replaced. If adenocarcinoma oxaliplatin.If squamos cell carcinoma carboplatin.
Radiation: Radiochemotherapy — Cisplantin 100 mg/m2 day 1. 5-fluoracil 750 mg/m2/24 hours infusion day 1-5. Three cycles. In the chemoradiation arm the radiotherapy start week 4 and continuing until week 7. Dose adjustet according to current LPK and TPK values.
  Other Names: Suffering moderate/severe hearing impairment and/or tinnitus cisplatin can be replaced. If adenocarcinoma oxaliplatin.If squamos cell carcinoma carboplatin.
  Arms: Radiochemotherapy

SUMMARY:
The purpose of this randomized study is to clarify if neoadjuvant radiochemotherapy gives a higher degree of complete histological response than neoadjuvant chemotherapy before surgery in patients undergoing treatment for cancer of the esophagus or cardia.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified squamos cell carcinoma, adenocarcinoma of the esopohagus or gastric cardia (type II)
* Tumor located in cervical oesophagus, not requiring laryngo-esophagectomy. Patients with performance status 0-1 axxording to WHO scale and with resectable tumours, as assessed at the prerandomisation evaluation
* Adequate haemotological function, defined as having WBC > 3 x 10(9)/litre and platelets > 100 x 10 (9)/litre.
* Adequate renal function defined as having normal serum creatinine level and/or calculated glomerular filtration rate > 60 ml/min.
* Tumour stage: T1Ni, T2N0, T2N1, T3N0, T3N1, M1a

Exclusion Criteria:

* Pregnancy and/or lactation. Women of childbearing ages can be included and provided that adequate contraceptive methods are used
* Patients with diabetes complications (e.g. rethinopathy, neuropathy) as well as patients with uncontrolled cardiac disease or myocard infarction within 12 months are considered unsuitable for chemoradiotherapy.
* Concomitant malignancy (< 5 years since diagnosis) that can interfere the interpretation of study results, ongoing antitumoral treatment.
* Patients being unable tom comply with the protocol
* Tumor stage T1 N0, T4 NX or TXNXM1b

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2018-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Nilsson, Professor, Principal Investigator — Karolinska University Hospital, Gastrocentrum; Lars Lundell, Professor, Study Chair — Karolinska University Hospital, Gastrocentrum
Locations (1):
- Upper Digestive Diseases. Department of surgery, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Klevebro F, Alexandersson von Dobeln G, Wang N, Johnsen G, Jacobsen AB, Friesland S, Hatlevoll I, Glenjen NI, Lind P, Tsai JA, Lundell L, Nilsson M. A randomized clinical trial of neoadjuvant chemotherapy versus neoadjuvant chemoradiotherapy for cancer of the oesophagus or gastro-oesophageal junction. Ann Oncol. 2016 Apr;27(4):660-7. doi: 10.1093/annonc/mdw010. Epub 2016 Jan 17. PMID 26782957
- [Result] Sunde B, Klevebro F, Johar A, Johnsen G, Jacobsen AB, Glenjen NI, Friesland S, Lindblad M, Ajengui A, Lundell L, Lagergren P, Nilsson M. Health-related quality of life in a randomized trial of neoadjuvant chemotherapy or chemoradiotherapy plus surgery in patients with oesophageal cancer (NeoRes trial). Br J Surg. 2019 Oct;106(11):1452-1463. doi: 10.1002/bjs.11246. Epub 2019 Aug 22. PMID 31436322
- [Result] von Dobeln GA, Klevebro F, Jacobsen AB, Johannessen HO, Nielsen NH, Johnsen G, Hatlevoll I, Glenjen NI, Friesland S, Lundell L, Yu J, Nilsson M. Neoadjuvant chemotherapy versus neoadjuvant chemoradiotherapy for cancer of the esophagus or gastroesophageal junction: long-term results of a randomized clinical trial. Dis Esophagus. 2019 Feb 1;32(2). doi: 10.1093/dote/doy078. PMID 30137281
- [Result] Klevebro F, Johnsen G, Johnson E, Viste A, Myrnas T, Szabo E, Jacobsen AB, Friesland S, Tsai JA, Persson S, Lindblad M, Lundell L, Nilsson M. Morbidity and mortality after surgery for cancer of the oesophagus and gastro-oesophageal junction: A randomized clinical trial of neoadjuvant chemotherapy vs. neoadjuvant chemoradiation. Eur J Surg Oncol. 2015 Jul;41(7):920-6. doi: 10.1016/j.ejso.2015.03.226. Epub 2015 Apr 8. PMID 25908010
- [Result] Sunde B, Johnsen G, Jacobsen AB, Glenjen NI, Friesland S, Lindblad M, Rouvelas I, Wang N, Lundell L, Lagergren P, Nilsson M. Effects of neoadjuvant chemoradiotherapy vs chemotherapy alone on the relief of dysphagia in esophageal cancer patients: secondary endpoint analysis in a randomized trial. Dis Esophagus. 2019 Feb 1;32(2). doi: 10.1093/dote/doy069. PMID 30084992
- [Derived] Lund M, Tsai JA, Nilsson M, Winter R, Lundell L, Kalman S. Effects of neoadjuvant chemo or chemoradiotherapy for oesophageal cancer on perioperative haemodynamics: A prospective cohort study within a randomised clinical trial. Eur J Anaesthesiol. 2016 Sep;33(9):653-61. doi: 10.1097/EJA.0000000000000480. PMID 27254026
- [Derived] Lund M, Alexandersson von Dobeln G, Nilsson M, Winter R, Lundell L, Tsai JA, Kalman S. Effects on heart function of neoadjuvant chemotherapy and chemoradiotherapy in patients with cancer in the esophagus or gastroesophageal junction - a prospective cohort pilot study within a randomized clinical trial. Radiat Oncol. 2015 Jan 13;10:16. doi: 10.1186/s13014-014-0310-7. PMID 25582305

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiochemotherapy: Radiochemotherapy + Surgery
  Radiochemotherapy: Cisplantin 100 mg/m2 day 1. 5-fluoracil 750 mg/m2/24 hours infusion day 1-5. Three cycles. In the chemoradiation arm the radiotherapy start week 4 and continuing until week 7. Dose adjustet according to current LPK and TPK values.
- Chemotherapy: Chemotherapy + surgery
  Chemotherapy: Cisplantin 100 mg/m2 day 1. 5-fluoracil 750 mg/m2/24 hours infusion day 1-5. Three cycles. In the chemoradiation arm the radiotherapy start week 4 and continuing until week 7. Dose adjustet according to current LPK and TPK values.
  Radiochemotherapy: Cisplantin 100 mg/m2 day 1. 5-fluoracil 750 mg/m2/24 hours infusion day 1-5. Three cycles. In the chemoradiation arm the radiotherapy start week 4 and continuing until week 7. Dose adjustet according to current LPK and TPK values.
Period: Overall Study
Arm/Group | Radiochemotherapy | Chemotherapy
Started | 90 | 91
Completed | 90 | 91
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: see Klevebro et al Annals of Oncology, primary outcome
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiochemotherapy | Chemotherapy | Total
Number analyzed (Participants) | 90 | 91 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 55 | 107
  >=65 years | 38 | 36 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 72 | 77 | 149
Region of Enrollment [Number; unit: participants]
  Sweden | 90 | 91 | 181

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Histological Response (pCR) After Resection Than Chemotherapy Alone in Patients With Resectable Carcinoma of the Esophagus and Cardia.
Description: Chireac tumour regression grade
Time Frame: Therapy followed in 14-16 weeks before surgery. After surgery the patients will be followed until 60 weeks after completed therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiochemotherapy | Chemotherapy
Number analyzed (Participants) | 78 | 78
Participants | 22 | 7

2. Secondary Outcome: Safety of Respective Neoadjuvant Therapies.
Description: Safety profile of carrying out radical surgery after respective neoadjuvant therapy.
Time Frame: Five years follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Radiochemotherapy | Chemotherapy
Number analyzed (Participants) | 90 | 91
Participants | 79 | 81

3. Secondary Outcome: HRQOL and Swallowing Function
Description: The European Organisation for Research and Treatment of Cancer (EORTC) core questionnaire QLQ-C30 and disease specific questionnaires (QLQ-OES24/OG25). All items included in the questionnaires are analysed and also separate analysis of dysphagia questionnaires for oesophageal cancer were used, both clinically and psychometrically validated. All questions have four response alternatives (1, not at all; 2:a little, 3: quite a bit, 4: very much), except global scales which comprise seven response alternatives from poor to excellent. Questionnaire responses were transformed lineraly into scores ranging from 0 to 100 according to the EORTC scoring manual. A higher score indicates either more symotoms or better function, depending on the question.
Time Frame: Entry study up to Five years follow up
Population: Number of patients who responded to quality of Life instruments the EORTC QLQ-C30 and the oesophageal specific instrument
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Radiochemotherapy | Chemotherapy
Number analyzed (Participants) | 80 | 74
units on a scale
  Mean global QoL | 67 [62 to 72] | 69 [63 to 74]
  Dysphagia score all | 27 [20 to 34] | 31 [24 to 39]

ADVERSE EVENTS:
Arm/Group | Radiochemotherapy | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 57/90 | 41/91
Other Adverse Events (participants affected / at risk) | 0/90 | 0/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiochemotherapy (N=90) | Chemotherapy (N=91)
SAE (Investigations) | 57 (57) | 41 (41)
Infection (Infections and infestations) | 5 (5) | 5 (5)
Nausea and vomiting (Gastrointestinal disorders) | 6 (6) | 2 (2)
Nutritional deficiency (Metabolism and nutrition disorders) | 13 (13) | 13 (13)
Gastrointestinal symptoms (Gastrointestinal disorders) | 5 (5) | 1 (1)
Cardiovascular events (Cardiac disorders) | 14 (14) | 7 (7)
Renal failure (Renal and urinary disorders) | 4 (4) | 7 (7)
Neutropenia/thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Other (General disorders) | 3 (3) | 3 (3)
Death (Cardiac disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No